CLINICAL TRIAL: NCT01608919
Title: Predictive Value of Whole Blood Coagulation Parameters for Post-discharge Venous Thromboembolism After Cancer Resection.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sara Cheng, MD has left the University of Colorado and we have closed this study.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-1295
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- diagnostic blood tests (No Intervention): We are using 2 standard approved blood tests that may be useful in predicting who may develop a venous thromboembolism after cancer surgery.
  Interventions: Other: blood tests

INTERVENTIONS:
Other: blood tests — thromboelastogram platelet mapping

SUMMARY:
This study plans to learn more about the role of 2 blood tests in predicting who might develop a blood clot in their arm or leg after major surgery. The investigators know that patients who have cancer and major surgery have a higher than normal risk of getting blood clots in the veins of their arms or legs. This can be very dangerous because the clot can move into your lungs.

DETAILED DESCRIPTION:
Venous Thromboembolism (VTE) after cancer surgery hospitalization is the most common cause of death at 30 days after cancer surgery, and is a significant source of patient morbidity and health care cost. Pharmacoprophylaxis has proven efficacy in preventing post-discharge VTE in surgical cancer patients, but perceived risks and costs pose barriers to widespread adoption by clinicians. Risk stratification of this patient population is necessary to allow appropriate prescription of prophylaxis to the highest risk patients. Can the investigators develop a risk stratification model that includes a readily available laboratory test, the thromboelastogram with or without platelet mapping?

ELIGIBILITY:
Inclusion Criteria:

* subjects who are having primary, open resection surgery of gastrointestinal or bladder cancer

Exclusion Criteria:

* currently receiving anticoagulation therapy
* pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolism free survival after surgery for gastrointestinal or urologic cancer | 3 months post-discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Sara Cheng, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States